CLINICAL TRIAL: NCT07275762
Title: A Multicenter, Randomized, Double-blind, Double-dummy, Parallel-controlled Phase II Clinical Study Evaluating the Efficacy and Safety of Y-4 Tablets in Chinese Patients With Postherpetic Neuralgia, Compared With Pregabalin Capsules
Brief Title: Y-4 to Treat the Postherpetic Neuralgia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Neurodawn Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Y-4-LC-04
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Postherpetic Neuralgia; Y-4; Pregabalin
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Y-4 group (Experimental): participants in this group will use pregabalin and riluzole
  Interventions: Drug: Y-4 tables
- pregabalin group (Other): participants in this group will use pregabalin only
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Y-4 tables — combination of pregabalin and riluzole
  Arms: Y-4 group
Drug: Pregabalin — only use pregabalin
  Arms: pregabalin group

SUMMARY:
The goal of this clinical trial is to assess the efficacy and safety of Y-4 in patients with postherpetic neuralgia(PHN).

The main questions it aims to answer are:

The efficacy of Y-4 to treat PHN. If drug RK-4 is safe and tolerate in the patients with LHI?

Researchers will analyze data from different groups, includes Y-4 group and pregabalin group , to see efficacy of Y-4 and If drug Y-4 is safe and tolerate in the patients with PHN.

Participants will :

* Take Y-4 (1w titration period:75 mg pregabalin +18.5 mg riluzole, 12w fixed dose period: 150 mg pregabalin +37.5 mg riluzole, 1w drug withdraw period: 1w titration period:75 mg pregabalin +18.5 mg riluzole) or pregabalin(75 mg for 1w titration period , 150 mg for 12w fixed dose period ,75 mg for 1w drug withdraw period) twice a day for 14 weeks after run-in period (placebo) lasting for 1 week.
* Visit the hospital according to the follow-up schedule agreed upon with your doctor. contact the research staff as soon as possible to reschedule when unable to attend the scheduled study visit.
* Use investigational products as directed by the doctor and undergo the related treatment.
* Inform their investigators of any changes in their health, including any side effects or symptoms, whether or not they believe these changes are related to the trial medication, as well as any new medications they are using or wish to use, or any changes in the dosage of medications they have already taking.
* Use reliable contraceptive methods , such as abstinence, intrauterine devices, double barrier methods (e.g., condom with spermicide or condom with a diaphragm containing spermicide), contraceptive implants, or oral contraceptives (except if the partner is infertile) during the study period and within one month after the study is completed.
* Must inform investigators immediately if they or their partner become pregnant during the study.
* Be sure to inform other doctors being consultant that you are participating in this clinical study.
* Restrict medication use and treatment during the study.

ELIGIBILITY:
Inclusion Criteria:

- 1. Able to understand and voluntarily sign the informed consent form. 2. Age ≥ 18 years, any gender. 3. Diagnosed with PHN, meaning pain persists for more than one month after the acute shingles rash has healed.

4. VAS score in SF-MPQ ≥ 40 mm of the last 24 hours during screening.

Exclusion Criteria:

* 1. Known previous allergy to the investigational products, rescue medication ingredients, other chemically similar drugs, or excipients.

  2. During screening, individuals who have been clearly diagnosed with peripheral neuropathy or pain unrelated to PHN (including but not limited to those caused by cerebrovascular disease, Guillain-Barré syndrome, cervical or lumbar spine disorders, osteoarticular or tendon lesions, chronic kidney disease or uremia, thyroid disease, intracranial tumors, trauma, etc.) and are judged by the investigator to potentially confound the assessment of PHN.

  3. During screen, suffer from a systemic disease that, in the opinion of the investigator, may affect the patient's participation in the study or affect the evaluation of the efficacy of PHN, including but not limited to:
  1. Severe cardiopulmonary diseases, such as unstable angina, myocardial infarction, severe arrhythmia within 6 months prior to screening, NYHA cardiac function classification of grade III~IV at screening, hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg at screening), recurrent asthma attacks, etc.;
  2. Chronic digestive diseases, such as liver fibrosis, chronic active hepatitis, peptic ulcer, etc.;
  3. Neuropsychiatric disorders, including epilepsy, recurrent dizziness or headache, cognitive impairment; Cerebrovascular disease (such as cerebral infarction) or recurrent transient ischemic attack within 6 months prior to screening;
  4. History of malignant tumors within 5 years prior to screening (excluding cured basal cell carcinoma of the skin, carcinoma in situ and papillary thyroid carcinoma);
  5. Presence of active infection, which, in the opinion of the investigator, is not suitable for entry into this study;
  6. Diabetic patients with poor glycemic control (peritoneal venous blood glucose ≥11mmol/L at screening);
  7. Suffering from immunocompromised diseases, such as systemic lupus erythematosus, acquired immunodeficiency syndrome, immunosuppressant therapy for autoimmune diseases.

  4. During screening, situations may exist that investigators believe could affect pain assessment, such as if the affected skin area has a skin condition that may influence sensation.

  5. Previously received nerve destruction for PHN, or underwent minimally invasive interventions (such as nerve blocks or neurostimulation), physical therapy (such as red light therapy), or traditional Chinese external treatments (such as acupuncture) within one week prior to screening.

  6. Use prohibited drugs within the first 5 half-lives, or change the restricted drug dosage within the first 14 days.

  7. Severe hematological, hepatatological, and renal function abnormalities at the time of screening, which meet any of the following laboratory test results: 1) Hematology: neutrophil count < 1.5×109/L, or platelet < 90×109/L, or hemoglobin <100g/L; 2) Liver function: ALT or AST > 2.5 times ULN; or TBIL > 1.5 times ULN; 3) Renal function: CrCL<60 mL/min/1.73 m2 (calculated based on Cockroft-Gault formula a); 4) Creatine kinase >2-fold ULN.

  8. Participants already diagnosed with sleep apnea, or those with severe snoring and daytime sleepiness, as well as intermittent hypoxia.

  9. Participants with a history of suicidal behavior, or those assessed to have suicidal tendencies using the Columbia-Suicide Severity Rating Scale (C-SSRS).

  10.Hepatitis B surface antigen (HBsAg) positive and HBV-DNA titer >lower limit of reference value, or hepatitis C virus antibody (HCV-Ab) positive and HCV-DNA titer >lower limit of reference value, or human immunodeficiency virus antibody (HIV-Ab) positive, or serum Treponema pallidum-specific antibodies (TP-Ab) positiv eand rapid plasma reagin/toluidine red unheated serum test (RPR or TRUST) positive at screening.

  11. Known drug abuse, or history of alcohol abuse within 1 year prior to screening, i.e., drinking more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of spirits with 40% alcohol or 150 mL of wine).

  12. Pregnant or lactating females. 13.Male (or their partner) or female subjects have a fertility plan during the whole study period and within 1 month after the end of the study or are unwilling to take one or more non-drug contraceptive measures (such as condoms, intrauterine devices, etc.) during the study period.

  14.Prior participation in any other clinical study of any other drug within 30 days prior to screening.

  15.Engaging in high-altitude work, driving motor vehicles, or operating heavy machinery with associated risks during the study period.

  16.Other conditions that are considered unsuitable by the investigator to participate in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of Y-4 in patients with PHN by Change from baseline in Average Daily Pain Score (ADPS) for each group at week 13. | week 13
  The average daily pain score is a commonly used clinical method for pain assessment. It converts the intensity of pain into numerical values (generally 0-10 points) based on patient self-reports or standardized scales. After recording multiple pain scores each day, an average is calculated to monitor changes in pain and treatment effects dynamically. The core function of pain scoring is to quantify the subjective experience of pain, helping doctors understand the degree of pain and adjust treatment plans. Commonly used scales include: Numeric Rating Scale (NRS): 0 points (no pain) to 10 points (worst pain imaginable).

SECONDARY OUTCOMES:
Evaluate the efficacy of Y-4 in patients with PHN by ADPS response rate (i.e., proportion of patients with a ≥ 30% and ≥ 50% decrease in ADPS from baseline) at week 13 | week 13
  The average daily pain score is a commonly used clinical method for pain assessment. It converts the intensity of pain into numerical values (generally 0-10 points) based on patient self-reports or standardized scales. After recording multiple pain scores each day, an average is calculated to monitor changes in pain and treatment effects dynamically. The core function of pain scoring is to quantify the subjective experience of pain, helping doctors understand the degree of pain and adjust treatment plans. Commonly used scales include: Numeric Rating Scale (NRS): 0 points (no pain) to 10 points (worst pain imaginable).
Evaluate the efficacy of Y-4 in patients with PHN by Change from baseline in Average Daily Pain Score (ADPS) for each group at week 1-12 and 14. | week 1-12 and 14
  The average daily pain score is a commonly used clinical method for pain assessment. It converts the intensity of pain into numerical values (generally 0-10 points) based on patient self-reports or standardized scales. After recording multiple pain scores each day, an average is calculated to monitor changes in pain and treatment effects dynamically. The core function of pain scoring is to quantify the subjective experience of pain, helping doctors understand the degree of pain and adjust treatment plans. Commonly used scales include: Numeric Rating Scale (NRS): 0 points (no pain) to 10 points (worst pain imaginable).
Evaluate the efficacy of Y-4 in patients with PHN by Change from baseline in Score of Average Daily Sleep Interference Score (ADSIS) in each group at week 1-14; | week 1-14
  The subject will select the number that best describes his or her sleep interference experience during the past 24 hours on a scale of 0 (pain did not interfere with sleep) to 10 (pain completely interfered with sleep)
Evaluate the efficacy of Y-4 in patients with PHN by The proportion of patients grading ≤2 and ≤3 in each group using Patient Global Impression of Change scale (PGIC) at week 1, 3, 5, 7, 11, 13, 14. | week 1, 3, 5, 7, 11, 13, 14
  The items of PGIC are listed as follows Score PGIC
  1. Very much improved
  2. Much improved
  3. Minimally improved
  4. No change
  5. Worse
  6. Much worse
  7. Very much worse
Evaluate the efficacy of Y-4 in patients with PHN by Change from baseline in Simplified McGill Pain Questionnaire (SF-MPQ) in each group at week 1, 3, 5, 7, 9, 11, 13, 14 (single score and total score); | week 1, 3, 5, 7, 9, 11, 13, 14
  The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors.(Throbbing, Shooting, Stabbing, Sharp, Cramping, Gnawing, Hot-burning, Aching, Heavy, Tender, Splitting, Tiring-exhausting, sickening, Fearful, Punishing-cruel)
Evaluate the efficacy of Y-4 in patients with PHN by Change from baseline in Hospital Anxiety and Depression Scale (HADS) at week 1, 3, 5, 7, 9, 11, 13, 14 | week 1, 3, 5, 7, 9, 11, 13, 14
  The Hospital Anxiety and Depression Scale (HADS) is a psychological assessment tool used to screen for anxiety and depression in patients at general hospitals. It was first developed by Zigmond and Snaith in 1983. The scale contains 14 items, divided into two subscales: anxiety (A) and depression (D), each consisting of 7 questions. Each item is scored on a 4-point scale from 0 to 3, with the total score for each subscale ranging from 0 to 21. Scores of 0-7 indicate no symptoms, 8-10 suggest possible symptoms, and 11-21 indicate definite symptoms. HADS was designed to avoid the use of indicators affected by physical illnesses and is suitable for screening psychological issues in patients with chronic diseases.
Evaluate the efficacy of Y-4 in patients with PHN by The amount of rescue medication acetaminophen tablets used by each group during the trial | the whole study（16 week）
  4-6 h per time, The maximum daily dose should not exceed 2.0 g, and continuous use should not exceed 5 days.
Evaluate the safety of Y-4 in patients with PHN by The incidence of treatment-emergent adverse events (TEAE) in each group. | the whole study(16 week)
  An AE is defined as any untoward medical event that occurs after receiving a drug or treatment or any deterioration of a disease or symptom that existed before receiving the investigational product or treatment (excluding the disease studied in this trial) in a subject or a clinical investigation subject, whether or not considered related to the investigational product or treatment. Therefore, an AE can be a discomfort sign (including an abnormal laboratory finding), symptom, or transient disease beyond any indication, whether or not related to the investigational product or treatment.
  The investigator will name each AE reported during the study by MedDRA PT and evaluate their severity using the criteria of CTCAE 5.0.
  The relevance evaluation is divided into 5 grades: 1-certainly related; 2-probably/likely related; 3-possibly related; 4-unlikely related; 5 not related.
Evaluate the safety of Y-4 in patients with PHN by rates of Significant Adverse Events. | the whole study(16 week)
  Significant Adverse Events refers to any adverse event, other than a serious adverse event, that leads to the implementation of targeted medical measures (such as drug withdrawal, dose reduction, and symptomatic treatment) and is significant in blood or other laboratory tests.
Evaluate the safety of Y-4 in patients with PHN by rates of Serious Adverse Events (SAE) after treatment. | the whole study(16 week)
  Serious Adverse Events (SAE) refers to adverse medical events that occur after a subject receives the investigational products, including death, life-threatening conditions, permanent or severe disability or functional loss, the subject requiring hospitalization or an extension of hospital stay, as well as congenital anomalies or birth defects.
Evaluate the safety of Y-4 in patients with PHN by incidence of subject getting abnormal results of vital signs after treatment. | the whole study(16 week)
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Vital signs(blood pressure, respiration, pulse, body temperature will be assessed by according equipments.(electronic sphygmomanometer thermometer).
Evaluate the safety of Y-4 in patients with PHN by incidence of subject getting abnormal results of physical examinations after treatment. | the whole study(16 week)
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Physical examinations will be conduct by the investigator through observation
Evaluate the safety of Y-4 in patients with PHN by incidence of subject getting abnormal results of 12-lead ECG after treatment. | the whole study(16 week)
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. 12-lead ECG will be analyzed by single RR Heart Rate, aggregate PR Interval, aggregate QRS Duration, aggregate RR Interval, aggregate QT Interval, aggregate QTC Interval. Normal range is provided by the site.
Evaluate the safety of Y-4 in patients with PHN by incidence of subject getting abnormal results of laboratory tests after treatment. | the whole study (16 week)
  Record changes from baseline to post-treatment, listing deviations from normal ranges post-treatment. Laboratory tests are composed of hematology, urinalysis, serum chemistry, coagulation test. Normal range is provided by the site.

IPD SHARING:
Plan to Share IPD: No